CLINICAL TRIAL: NCT02747342
Title: A Phase 1 Trial of SHR3680 With or Without SHR3162 in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase 1 Trial of SHR3680 With or Without SHR3162 in Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-002
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Neoplasm; Prostate Cancer
Keywords: Metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR3680; SHR3680+SHR3162 (Experimental): In dose esclation and expansion phase, SHR3680 will be administered orally In combination phase, SHR3680 will be administered together with SHR3162
  Interventions: Drug: SHR3680; SHR3162

INTERVENTIONS:
Drug: SHR3680; SHR3162 — SHR3680 will be administered orally in dose escalation/expansion phase,
  SHR3680 will be administered orally at a fixed dose together with SHR3162 in combination phase.

SUMMARY:
This is a multicenter, dose-escalation/expansion phase 1 trial to evaluate the safety, tolerability and efficacy of SHR3680 with or without SHR3162 given orally to subjects with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This study consists of 2 Part. In the Part 1 (dose escalation phase), up to 4 dose levels of SHR3680 will be investigated with a sequential "3+3" design (3 or 6 participants in each dose level). There will be a single-dose pharmacokinetic (PK) run-in period (7 days). Following the first dose, participants will enter a 1 week treatment-free period to evaluate safety and single-dose PK. If not dose-limiting toxicities (DLTs) are observed during the 1-week period, SHR3680 administration will resume at the same dose level.

In the Part 2a (expansion phase), up to 9 additional participants will be enrolled at the MTD or recommended phase 2 dose (RP2D). The purpose of the expansion part of the study is to explore the clinical benefits of SHR3680 and to further identify its PK features.

In Part 2b (combination phase), two dose cohorts of SHR3162 combine with SHR3680 at fixed dose will be investigated.

ELIGIBILITY:
Inclusion Criteria

1. Male 18 years and older
2. Ability to understand the purposes and risks of the trial and his/her signed informed consent form approved by the HREC of the trial site, which must be obtained before entering the trial
3. Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
4. For patients who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the trial
5. Serum testosterone level < 1.7 nmol/L (50 ng/dL) at the screening visit
6. Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration)
7. Progressive disease by PSA or imaging after docetaxel-based chemotherapy or abiraterone in the setting of medical or surgical castration. Prior enzalutamide is allowed as long as patients had a PSA response >50% or were treated for at least 6 months. Disease progression for study entry is defined by one or more of the following three criteria:

   * PSA progression defined by a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the Screening visit should be ≥2 μg/L (2 ng/mL)
   * Soft tissue disease progression defined by RECIST (Appendix A)
   * Bone disease progression defined by two or more new lesions on the bone scan
8. ECOG performance status of 0 or 1
9. Life expectancy of at least 6 months
10. Able to swallow the study drug and comply with study requirements
11. Acceptable liver function defined as:

    * Total bilirubin ≤ 1.5 times the upper limit of normal range (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN; however, ≤ 5 times ULN in a subject who has liver metastases or has been treated with biliary drainage
12. Acceptable renal function defined below:

    • Serum creatinine ≤ 1.5 times ULN
13. Acceptable hematologic status (without hematologic support including hematopoietic factor, blood transfusion) defined below:

    * Absolute neutrophil count (ANC) ≥ 1,500/μL
    * Platelet count ≥ 100,000/μL
    * Hemoglobin ≥ 9.0 g/dL

Exclusion Criteria

1. Treatment with AR antagonists (enzalutamide, bicalutamide, flutamide, nilutamide), 5-α reductase inhibitors (finasteride, dutasteride), estrogens, or chemotherapy within 4 weeks of enrollment (day 1 visit) or plans to initiate treatment with any of these drugs during the study. Ongoing therapy with bisphosphonates or Rank Ligand inhibitors are acceptable.
2. Prior treatment with a PARP inhibitor or have plans to initiate treatment with a PARP inhibitor during the study (only apply to subjects participating in Part 2b)
3. Treatment with therapeutic immunizations for prostate cancer (e.g., PROVENGE®) or plans to initiate treatment with any of these therapies during the study
4. Metastases in the brain or active epidural disease (Note: patients with treated for epidural disease are allowed to enter the trial)
5. Use of herbal products that may decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within 4 weeks of enrollment (day 1 visit) or plans to initiate treatment with any of these therapies during the study
6. History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer
7. Radiation therapy within 3 weeks (if single fraction of radiotherapy, then a 1-week gap is allowable) and radionuclide therapy within 8 weeks of enrollment (Day 1 visit). Any radiotherapy-related AE > Grade 1 before the start of study treatment.
8. Have used or plan to use from 30 days prior to enrollment (day 1 visit) through to the end of the study medications known to lower the seizure threshold or prolong the QT-interval (described in Appendix I)
9. Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular disease
10. Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment
11. History of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attack within 12 months of enrollment (day 1 visit), or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization)
12. Use of an investigational agent within 4 weeks of enrollment or plans to initiate treatment with an investigational agent during the study
13. Major surgery, other than diagnostic surgery, within 4 weeks prior to trial entry, without complete recovery
14. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within the last 3 months)
15. Structurally unstable bone lesions suggesting impending fracture

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 4 weeks
  MTD is defined as the maximum dose level at which no more than 1 out of 3 participants experience a DLT within the first 4 weeks of multiple dosing
Recommended Phase 2 doses (RP2Ds) | 24 months
  RP2D will be determined based on the available data for toxicity and PK.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | 24 months
  The number and proportion of subjects experiencing treatment-emergent AEs (TEAE); drug exposure; clinically significant changes in laboratory parameters, vital signs, physical examinations, weight, ECOG performance status, ECG abnormalities, number and causes of deaths.
The AUC of SHR3680 and SHR3162 (area under the curve) | 4 weeks
  The AUC of SHR3680 given as BID 240 mg tablets in combination with SHR3162
The cMax (peak plasma concentration) of SHR3680 and SHR3162 | 4 weeks
  The cMax (peak plasma concentration) of SHR3680 given as BID 240 mg tablets in combination with SHR3162
PSA reduction | 12 weeks
  Percentage of participants reaching at least a 50% reduction in prostate specific antigen (PSA) at Week 12 as compared to baseline
PSA progression | 24 months
  Time to reach the PSA Progression
Objective response rate (ORR) | 24 months
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time periodthe proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
Radiological progression-free survival (PFS) | 24 months
  the length of time during and after the treatment

OTHER OUTCOMES:
Homologous recombination deficiency (HRD) | 2 weeks
  Homologous recombination deficiency (HRD) as a predictive biomarker of response in patients with Metastatic castration resistant prostate cancer

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Border Medical Oncology, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Icon Cancer Centre, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No